CLINICAL TRIAL: NCT06025487
Title: Immunogenicity and Safety of a Meningococcal Serogroup B Vaccine in Adult Patients with Asplenia
Brief Title: Meningococcal B Vaccine in Patients with Asplenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nicole Harrison, Dr. Nicole Harrison, Consultant for Infectious Diseases and Tropical Medicine, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MenB_Asplenia; 2022-001451-16 (EudraCT Number)
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Splenectomy; Status
Keywords: Asplenia; Meningococcal disease; Meningococcal B vaccine
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine

STUDY DESIGN:
Intervention Model Description: prospective open-label phase II study comparing patients and healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Active Comparator): Asplenic patients receiving two doses of Bexsero (meningococcal B vaccine) with one-month interval between doses
  Interventions: Biological: Bexsero
- Healthy controls (Active Comparator): Healthy controls receiving two doses of Bexsero (meningococcal B vaccine) with one-month interval between doses
  Interventions: Biological: Bexsero

INTERVENTIONS:
Biological: Bexsero — two doses of Bexsero are applied intramuscularly with a one-month interval between doses

SUMMARY:
Patients without a spleen (asplenia) experience an increased risk for septicaemia from encapsulated bacteria, which is associated with a high mortality rate. Meningococcal bacteria can cause such infections and serogroup B is the dominant meningococcal subtype in Europe. Therefore, vaccination for risk populations like patients without a spleen is a pressing matter. Considering the effectiveness of the meningococcal serogroup B vaccine, data for this high-at-risk population is currently lacking. The aim of this study is to evaluate the meningococcal B vaccine (BEXSERO®) in patients without a spleen compared to a healthy control group. A total of 40 patients and 40 healthy persons will receive a two-dose schedule of BEXSERO® with a one-month interval between doses. The effectiveness of the vaccine will be determined by measuring antibodies against different meningococcal strains in the blood of the patient. The amount of antibodies one month after second vaccination will be compared between patients and healthy persons. The most reliable assay to determine antibodies against meningococcal strains is the human serum bactericidal assay which will be carried out in a reference laboratory. Other end points are the persistence of antibodies after six months and the cellular immune response. The cellular immune response will be assessed by measuring the proliferation of certain immune cells like lymphocytes and the amount of produced cytokines (signalling proteins) after vaccination. In addition, the safety of the vaccine will be evaluated by documenting all adverse reactions to the vaccine. Overall, this study will be the first to assess the effectiveness of the meningococcal B vaccine in this high-at-risk population and provide data for vaccination guidelines.

DETAILED DESCRIPTION:
This study is a prospective open-label phase II pilot study to assess the immunogenicity and safety of BEXSERO® in asplenic patients. Patients participating in the study will complete a total of four study visits. A two dose schedule of BEXSERO® will be applied intramuscularly with a one month interval between doses. Seropositivity will be assessed at baseline during the first visit, one month and six months after the second vaccination. Basic demographic data (gender, age) and medical data (type of asplenia, time of splenectomy, underlying diseases, concurrent medical conditions, medication etc) will be entered into a case report form (CRF). During the second and third visit all adverse events will be entered into the CRF and severe adverse events (SAEs) will be reported accordingly. Patients who have either been splenectomised or suffer from functional asplenia will be recruited for this study during their routine vaccination visit at the out-patient ward for infectious diseases of the Medical University of Vienna. A total of 40 patients and 40 healthy controls will be recruited for this study. The null hypothesis states that the immunogenicity of the meningococcal B vaccine is inferior in asplenic patients compared to a healthy control group. Immunogenicity will be assessed by human serum bactericidal antibody assay (hSBA) against three vaccine antigens. The human serum bactericidal antibody assay (hSBA) will be carried out in a reference laboratory (Meningococcal Reference Unit, Health Protection Agency North West Laboratory, Manchester Royal Infirmary, United Kingdom) to determine functional antibodies against three meningococcal vaccine antigens: PorA (strain NZ98/254), fHbp (strain 44/76-SL) and NadA (strain 5/99). The hSBA measures complement mediated killing of Neisseria meningitidis by vaccine-induced antibodies. It is considered as the "gold standard" for measuring antibody response against meningococcal bacteria. Currently, the detection of antibodies by hSBA with a titre of ≥1:4 is considered as a correlate for protection against meningococcal disease. The primary end point is the mean log-titre over the three meningococcal strains (NZ98/254 for PorA, 5/99 for NadA and 44/76-SL for fHbp) as measured by the hSBA one month after second vaccination. The non-inferiority margin was set to a 2-fold titre difference between the geometric mean titre of the asplenic group and the healthy control group. To investigate cellular immunity following meningococcal vaccination, lymphocyte proliferation and cytokine detection assays will be used.

ELIGIBILITY:
Inclusion Criteria:

For asplenic patients:

* asplenia due to splenectomy or functional asplenia
* 18 to 60 years of age
* if female: have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study
* providing written informed consent

For healthy controls:

* 18 to 60 years of age
* if female: have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study
* providing written informed consent

Exclusion Criteria:

For asplenic patients:

* pregnant or lactating
* febrile illness within last two weeks prior to enrolment
* allergic reactions to vaccination in past
* chemotherapy with Rituximab within last six months or during study period
* more than 20mg prednisone per day within last four weeks prior or at the time of enrolment
* previous vaccination against meningococcal serogroup B

For healthy controls:

* pregnant or lactating
* febrile illness within last two weeks prior to enrolment
* allergic reactions to vaccination in past
* any immunosuppressive condition or medication
* previous vaccination against meningococcal serogroup B

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Humoral immunogenicity | one month after second vaccination
  Immunogenicity will be assessed by human serum bactericidal antibody assay (hSBA) against three vaccine antigens (PorA, fHbp and NadA). The primary end point is the mean log-titre over the three meningococcal strains (NZ98/254 for PorA, 5/99 for NadA and 44/76-SL for fHbp) as measured by the hSBA one month after second vaccination.
  The non-inferiority margin was set to a 2-fold titre difference between the geometric mean titre of the asplenic group and the healthy control group.

SECONDARY OUTCOMES:
Persistence of humoral immunity | six months after second vaccination
  The persistence of antibodies six months after second vaccination as measured by hSBA
Cellular immunogenicity - lymphocyte proliferation | one month after second vaccination
  The cellular immune response as measured by lymphocyte proliferation assay
Cellular Immunogenicity - cytokine levels | one month after second vaccination
  The cellular immune response as measured by cytokine levels using Luminex
Adverse Events | four weeks after first and second vaccination
  Evaluation of safety by documenting all adverse events after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harrison, Dr., Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No